CLINICAL TRIAL: NCT04901117
Title: Bismuth-containing Quadruple Therapy for Helicobacter Pylori Eradication: A Multicenter Randomized Clinical Trial of 10 and 14 Days
Brief Title: Bismuth-containing Quadruple Therapy for Helicobacter Pylori Eradication: A Randomized Clinical Trial of 10 and 14 Days
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); The People's Hospital of Guangrao (Unknown); Weihai Municipal Hospital (Other); Shandong Province Third hospital (Other); Taian City Central Hospital (Other); Jining No.2 People's Hospital (Unknown); Maternity and Child Care Health Center of Dezhou (Unknown); Zoucheng People's Hospital (Unknown); Heze Municipal 3rd people's hospital (Unknown); Yuncheng Chengxin Hospital (Unknown); Peking University Care Luzhong Hospital (Other); Qihe County City Hospital (Unknown); Weifang People's Hospital (Other); Qilu Hospital of Shandong University (Other); Shandong Electric Power Central Hospital (Unknown)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SDU-QILU-G001
Record Dates: First submitted 2021-05-24; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Bismuth-containing quadruple regimen
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Tetracycline; Metronidazole

STUDY DESIGN:
Intervention Model Description: This trial is a multi-center, open-label, non-inferiority, randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-day treatment group (Experimental): Use the following drug combination option for 10 days. Option 1: Amoxicillin + Clarithromycin + Bismuth + Vonoprazan fumarate Option 2: Amoxicillin + Tetracycline + Bismuth + Vonoprazan fumarate Option 3: Amoxicillin + Metronidazole + Bismuth + Vonoprazan fumarate Three options are selected according to the hospital's situation.
  The dosage of each drug is:
  Amoxicillin (Amoxicillin, United Laboratories Co., Ltd.) 1000mg bid Clarithromycin (Klacid, Abbott S.r.l) 500mg bid Tetracycline 500mg qid Metronidazole400mg qid Bismuth Potassium Citrate (Livzon Pharmaceutical Group Inc.) 220mg bid Colloidal Bismuth Pectin (North China Pharmaceutical Co., Ltd.) 200mg bid Vonoprazan fumarate (VOCINTI, Takeda Pharmaceutical Company Limited, Hikari Plant) 20mg bid
  Interventions: Drug: Amoxicillin; Drug: Clarithromycin; Drug: Tetracycline; Drug: Metronidazole; Drug: Bismuth Potassium Citrate; Drug: Colloidal Bismuth Pectin; Drug: Vonoprazan fumarate
- 14-day treatment group (Active Comparator): Use the following drug combination option for 14 days. Option 1: Amoxicillin + Clarithromycin + Bismuth + Vonoprazan fumarate Option 2: Amoxicillin + Tetracycline + Bismuth + Vonoprazan fumarate Option 3: Amoxicillin + Metronidazole + Bismuth + Vonoprazan fumarate Three options are selected according to the hospital's situation.
  The dosage of each drug is:
  Amoxicillin (Amoxicillin, United Laboratories Co., Ltd.) 1000mg bid Clarithromycin (Klacid, Abbott S.r.l) 500mg bid Tetracycline 500mg qid Metronidazole400mg qid Bismuth Potassium Citrate (Livzon Pharmaceutical Group Inc.) 220mg bid Colloidal Bismuth Pectin (North China Pharmaceutical Co., Ltd.) 200mg bid Vonoprazan fumarate (VOCINTI, Takeda Pharmaceutical Company Limited, Hikari Plant) 20mg bid
  Interventions: Drug: Amoxicillin; Drug: Clarithromycin; Drug: Tetracycline; Drug: Metronidazole; Drug: Bismuth Potassium Citrate; Drug: Colloidal Bismuth Pectin; Drug: Vonoprazan fumarate

INTERVENTIONS:
Drug: Amoxicillin — Use according to the drug combination options selected by each center.
Drug: Clarithromycin — Use according to the drug combination options selected by each center.
Drug: Tetracycline — Use according to the drug combination options selected by each center.
Drug: Metronidazole — Use according to the drug combination options selected by each center.
Drug: Bismuth Potassium Citrate — Use according to the drug combination options selected by each center.
Drug: Colloidal Bismuth Pectin — Use according to the drug combination options selected by each center.
Drug: Vonoprazan fumarate — Use according to the drug combination options selected by each center.

SUMMARY:
The researchers collect treatment-naive H.pylori-positive patients from the outpatient clinic. The subjects were randomized to receive a 10-day or 14-day course of quadruple eradication therapy. 6-8 weeks after treatment, the subjects will re-take the 13C-urea breath test. Calculate the eradication rates, adverse reaction rates, patient compliance and cost-effectiveness index of each group.

DETAILED DESCRIPTION:
The researchers collect treatment-naive H.pylori-positive patients from the outpatient clinic. If the subject meets the selection criteria but not the exclusion criteria, and signs an informed consent form, the researchers randomized the subjects in groups: subjects received a 10-day or 14-day course of bismuth-containing quadruple eradication therapy. The medication of groups are as follows. 6-8 weeks after the eradication treatment, the subjects will review the 13C-urea breath test, and the researcher records the results.

After all subjects were tested, the eradication rates, adverse reaction rates, patient compliance and cost-effectiveness index of each group were calculated.

According to the course of treatment, it is randomized into a 10-day treatment group and a 14-day treatment group. The two groups of bismuth quadruple regimens are the same, as follows:

Option 1: Amoxicillin + Clarithromycin + Bismuth + Vonoprazan fumarate Option 2: Amoxicillin + Tetracycline + Bismuth + Vonoprazan fumarate Option 3: Amoxicillin + Metronidazole + Bismuth + Vonoprazan fumarate Three options are selected according to the hospital's situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65.
* Patients with H.pylori infection (Positive for any of the following: H.pylori culture, histopathology test, rapid urease test, 13C/14C-urea breath test, stool H.pylori antigen test).
* Patients whose birth place and residence within five years of birth are Shandong Province.
* Patients who have never received H. pylori eradication treatment.

Exclusion Criteria:

* Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than 3 times the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.
* Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.
* Patients with active gastrointestinal bleeding.
* Patients with a history of upper gastrointestinal surgery.
* Patients allergic to treatment drugs.
* Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs within 4 weeks
* Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse
* Patients whose current residence is not in Shandong Province.
* Patients whose re-check 13C/14C-urea breath test is negative before the start of the test.
* Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | Immediately after follow-up check.
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after follow-up check.
  Rate of adverse reactions
Patient compliance | Immediately after follow-up check.
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.
Cost-effectiveness index | Immediately after follow-up check.
  Ratio of costs to effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China

REFERENCES:
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Background] Liu WZ, Xie Y, Lu H, Cheng H, Zeng ZR, Zhou LY, Chen Y, Wang JB, Du YQ, Lu NH; Chinese Society of Gastroenterology, Chinese Study Group on Helicobacter pylori and Peptic Ulcer. Fifth Chinese National Consensus Report on the management of Helicobacter pylori infection. Helicobacter. 2018 Apr;23(2):e12475. doi: 10.1111/hel.12475. Epub 2018 Mar 7. PMID 29512258
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Background] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546
- [Background] Dore MP, Farina V, Cuccu M, Mameli L, Massarelli G, Graham DY. Twice-a-day bismuth-containing quadruple therapy for Helicobacter pylori eradication: a randomized trial of 10 and 14 days. Helicobacter. 2011 Aug;16(4):295-300. doi: 10.1111/j.1523-5378.2011.00857.x. PMID 21762269
- [Background] Rowland M, Daly L, Vaughan M, Higgins A, Bourke B, Drumm B. Age-specific incidence of Helicobacter pylori. Gastroenterology. 2006 Jan;130(1):65-72; quiz 211. doi: 10.1053/j.gastro.2005.11.004. PMID 16401469
- [Background] O'Ryan ML, Rabello M, Cortes H, Lucero Y, Pena A, Torres JP. Dynamics of Helicobacter pylori detection in stools during the first 5 years of life in Chile, a rapidly developing country. Pediatr Infect Dis J. 2013 Feb;32(2):99-103. doi: 10.1097/INF.0b013e318278b929. PMID 23076385
- [Background] Qiao C, Li Y, Liu J, Ji C, Qu J, Hu J, Ji R, Wan M, Lin B, Lin M, Qi Q, Zuo X, Li Y. Clarithromycin versus furazolidone for naive Helicobacter pylori infected patients in a high clarithromycin resistance area. J Gastroenterol Hepatol. 2021 Sep;36(9):2383-2388. doi: 10.1111/jgh.15468. Epub 2021 Mar 10. PMID 33691344